CLINICAL TRIAL: NCT01720758
Title: Assessment of the V600E Mutation in the B-RAF Gene in Chronic Lymphoproliferative Disease.
Acronym: B-RAF V600E
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: EMC-0124-11-CTIL
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Hairy Cell Leukemia; Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Leukemia, Hairy Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — perpheral blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The presence of a specific mutation in the gene known as B-RAF has been found in patients who have Hairy Cell Leukemia. In this study this specific mutation known as V600E will be ascertained in peripheral blood samples of patients who have this disease and in a group of patients who have a similar chronic lymphoproliferative conditions such as splenic marginal lymphoma. The finding of this specific mutation will help to verify or exclude the diagnosis of Hairy Cell Leukemia and determine whether patients are in remission.

ELIGIBILITY:
Inclusion Criteria:

Patients over the age of 18 years -

Exclusion Criteria:

Patients less than 18 years in age or mentally defectives.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are followed up in the Haematology Department in the Emek Medical Center for Hairy Cell Leukemia or chronic lymphoproliferative disease such as Splenic Marginal Zone Lymphoma. Patients who are examined and suspected to have Hairy Cell Leukemia.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
detection of the B-RAF V600E mutation | 2 weeks